CLINICAL TRIAL: NCT05265520
Title: His-Bundle Corrective Pacing in Heart Failure
Acronym: HIS-CRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Valentina Kutyifa, Associate Professor of Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY 00007025; 1R01HL153390-01A1 (NIH)
Record Dates: First submitted 2022-02-10; First posted 2022-03-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Right Bundle-Branch Block; Heart Failure; His-bundle Pacing; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Bundle-Branch Block; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- His-CRT implantation (Active Comparator): His-CRT implantation includes implantation of three leads, an endocardial right atrial lead, an endocardial right ventricular lead, and an endocardial His-bundle pacing leads directly pacing the intrinsic conduction system.
  Interventions: Procedure: His-CRT implantation
- BIV-CRT implantation (Active Comparator): BIV-CRT implantation includes implantation of three leads, an endocardial right atrial lead, an endocardial right ventricular lead, and an epicardial left ventricular lead implanted in a branch of the coronary sinus.
  Interventions: Procedure: BIV-CRT implantation

INTERVENTIONS:
Procedure: His-CRT implantation — The pathophysiological process is utilized in His-Bundle corrective pacing, resulting in a faster and more homogeneous activation of the heart pacing directly via the intrinsic conduction system of the heart accompanied by a right atrial endocardial lead and a right ventricular endocardial lead.
  Arms: His-CRT implantation
Procedure: BIV-CRT implantation — Biventricular cardiac resynchronization therapy has been shown to improve outcomes by delivering synchronized electrical stimuli to the right and left ventricles utilizing an an endocardial right atrial lead, an endocardial right ventricular lead, and an epicardial left ventricular lead implanted in a branch of the coronary sinus.
  Arms: BIV-CRT implantation

SUMMARY:
The investigators aim to prospectively evaluate the efficacy and mechanism of benefit of His-bundle pacing enhanced cardiac resynchronization therapy (His-CRT) vs. cardiac resynchronization therapy (BIV-CRT) in patients with heart failure and right bundle branch block (RBBB).

DETAILED DESCRIPTION:
In this prospective, randomized, multi-center clinical trial, the investigators aim to prospectively evaluate the efficacy and mechanism of benefit of His-bundle pacing enhanced cardiac resynchronization therapy (His-CRT) vs. cardiac resynchronization therapy (BIV-CRT) in patients with Right Bundle Branch Block (RBBB) Electrocardiogram (ECG) Pattern by assessing the improvement in left ventricular ejection fraction (LVEF) in the His-CRT vs. BIV-CRT arm at 6 months, and by evaluating changes in ECG biomarkers, NT-pro-brain natriuretic peptide (NT-proBNP) levels, and echocardiography biomarkers (left ventricular volumes, strain contractility, and dyssynchrony), as well as temporal changes in functional status and quality of life in the His-CRT vs. BIV-CRT arm at 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older (no upper age limit)
* Optimal medical therapy for heart failure by current guidelines
* Class IIa or IIb guideline-based indication for CRT-D implant in RBBB patients, including one of the following:

  * New York Heart Association (NYHA) class II HF symptoms, LVEF ≤ 30% and QRS≥ 150 ms (IIb); OR
  * NYHA class III-IV a HF, LVEF ≤ 35%, and QRS duration ≥ 150 ms (IIa); OR
  * NYHA class III-IV a HF, LVEF ≤ 35%, and QRS duration 120-149 ms (IIb)

Exclusion Criteria:

* Unable to obtain most recent imaging data from echocardiogram within 1 year prior to date of randomization
* Left bundle branch block (LBBB) or intraventricular conduction delay (IVCD) ECG morphology
* Unable or unwilling to follow study protocol
* Less than 12 months life expectancy at consent
* Pregnancy or planned pregnancy during duration of the study
* On heart transplant list or likely to undergo heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction at 6 months with His-CRT vs. BIV-CRT, in heart failure patients with Right bundle branch block (RBBB) | 6 month
  The effect of His-CRT vs. BIV-CRT on left ventricular ejection fraction (as a percentage) measured during an echocardiography imaging study will be analyzed using an analysis of covariance model for changes in LVEF from pre-implantation (baseline) to post-implantation (6 months follow-up), with randomized treatment group as the factor of interest, and baseline LVEF as a covariate. A t-test will be performed using this model to compare the adjusted group means, and a confidence interval will be constructed for their difference.

SECONDARY OUTCOMES:
Assess the mechanism of benefit with His-CRT vs. BIV-CRT by evaluating changes in ECG biomarkers | 6 months
  Secondary endpoint measured on a continuous scale of paced ventricular depolarization (QRS) duration in the His-CRT vs. BIV-CRT arm
Assess the mechanism of benefit with His-CRT vs. BIV-CRT by evaluating changes in echocardiographic left ventricular end-systolic volume (LVESV) | 6 months
  Secondary endpoint measured from echocardiography on left ventricular end-systolic volume (LVESV) in the His-CRT vs. BIV-CRT arm
Assess the mechanism of benefit with His-CRT vs. BIV-CRT by evaluating changes in echocardiographic left ventricular end-diastolic volume (LVEDV) | 6 months
  Secondary endpoint measured from echocardiography on left ventricular end-diastolic volume (LVEDV) in the His-CRT vs. BIV-CRT arm
Assess the mechanism of benefit with His-CRT vs. BIV-CRT by evaluating changes in NT-proBNP | 6 months
  Secondary endpoint of NT-proBNP in the His-CRT vs. BIV-CRT arm

OTHER OUTCOMES:
Ascertain the mechanism of benefit on ventricular depolarization (QRS duration) over time, at 6 months, 12 months, and 24 months. | Up to 24 months
  Assessing changes in QRS duration at 6, 12, 24 months in the His-CRT vs. BIV-CRT arm
Heart failure (HF) or death events | Up to 24 months
  Assess heart Failure (HF)/death rates in the His-CRT vs. BIV-CRT arm

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Kutyifa, MD, PhD, Principal Investigator — University of Rochester; Roderick Tung, MD, Principal Investigator — University of Arizona
Locations (14):
- United States (14):
  - University of Arizona, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of South Florida, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Valley Health System, Ridgewood, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Mission Health, Asheville, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - University of Vermont, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia